CLINICAL TRIAL: NCT00610012
Title: Clinical Registry Describing Treatment Reality and Therapy Modality of Patients With Metastatic or Locally Advanced Renal Cell Carcinoma Requiring Therapy
Brief Title: Tumor Registry of Advanced Renal Cell Carcinoma
Acronym: RCC-Registry
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitskreis Klinische Studien (Other); Bund der Urologen e.G. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOM RCC
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced Renal Cell Carcinoma; MRCC; Therapy-reality; Observation; Registry; RCC; ARCC; Germany; Metastatic Renal Cell Carcinoma; Renal Cell Carcinoma; Renal Cell Cancer; Sorafenib; Sunitinib; Interferon; Interleukin; Temsirolimus; Pazopanib; Cytokines; VEGF
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to record information of therapy reality of metastatic or locally advanced Renal Cell Carcinoma by office-based medical oncologists in Germany.

DETAILED DESCRIPTION:
The RCC Registry is a prospective, longitudinal, nation wide cohort study that collects data on the treatment reality of patients with mRCC. At inclusion, data in patient characteristics, comorbidities, tumor characteristics, and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented. Patients are followed until death or for a maximum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or locally advanced Renal Cell Carcinoma requiring therapy
* Start of first palliative therapy within 1 year before enrollment of patient to registry; since enrollment of 1000 Patients: start of first palliative therapy within 4 weeks before enrollment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Practitioners specialized in oncology and urology in Germany
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Documentation of therapies | 9 years, 3 years per patient

SECONDARY OUTCOMES:
Documentation of response rate and adverse reactions; development of a numeric prognostic score | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Goebell Peter, MD, Study Chair — Waldkrankenhaus St. Marien, Erlangen, Germany; Lothar Müller, MD, Study Chair — Onkologie Leer - Emden - Papenburg, Germany
Locations (1):
- iOMEDICO, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] P J G, A M, L M, H J H, M K, S B, N M. A cross-sectional investigation of fatigue in advanced renal cell carcinoma treatment: results from the FAMOUS study. Urol Oncol. 2014 Apr;32(3):362-70. doi: 10.1016/j.urolonc.2013.09.009. Epub 2013 Dec 8. PMID 24321255
- [Result] Goebell PJ, Muller L, Hurtz HJ, Koska M, Busies S, Marschner N. A Cross-Sectional Investigation of Fatigue, Mucositis, Hand-Foot Syndrome and Dysgeusia in Advanced Renal Cell Carcinoma Treatment: Final Results From the FAMOUS Study. Clin Genitourin Cancer. 2016 Feb;14(1):63-8. doi: 10.1016/j.clgc.2015.09.004. Epub 2015 Sep 25. PMID 26520429
- [Result] Marschner N, Staehler M, Muller L, Nusch A, Harde J, Koska M, Janicke M, Goebell PJ; RCC Registry Group. Survival of Patients With Advanced or Metastatic Renal Cell Carcinoma in Routine Practice Differs From That in Clinical Trials-Analyses From the German Clinical RCC Registry. Clin Genitourin Cancer. 2017 Apr;15(2):e209-e215. doi: 10.1016/j.clgc.2016.08.022. Epub 2016 Sep 8. PMID 27720164
- [Result] Goebell PJ, Staehler M, Muller L, Nusch A, Scheffler M, Sauer A, von Verschuer U, Tech S, Kruggel L, Janicke M, Marschner N; RCC-Registry Group (Tumour Registry of Advanced Renal Cell Carcinoma). Changes in Treatment Reality and Survival of Patients With Advanced Clear Cell Renal Cell Carcinoma - Analyses From the German Clinical RCC-Registry. Clin Genitourin Cancer. 2018 Dec;16(6):e1101-e1115. doi: 10.1016/j.clgc.2018.06.006. Epub 2018 Jun 27. PMID 30061035
- [Result] Goebell PJ, Muller L, Hubner A, Harich HD, Boller E, Koska M, Janicke M, Marschner N; RCC-Registry Group (Tumour Registry of Advanced Renal Cell Carcinoma). Body mass index as independent predictor of overall survival in patients with advanced renal cell carcinoma at start of systemic treatment-Analyses from the German clinical RCC-Registry. Urol Oncol. 2018 Oct;36(10):470.e1-470.e9. doi: 10.1016/j.urolonc.2018.07.007. Epub 2018 Aug 18. PMID 30131294
- [Result] Marschner N, Muller L, Munch A, Blumenstengel K, Hutzschenreuter U, Busies S. Adverse reactions in mRCC patients documented in routine practice by German office-based oncologists and uro-oncologists. J Oncol Pharm Pract. 2017 Jun;23(4):288-295. doi: 10.1177/1078155216632379. Epub 2016 Feb 22. PMID 26908232